CLINICAL TRIAL: NCT01865695
Title: Randomized, Double Blind, Placebo-controlled Trial of Creon in Patients With Low Faecal Pancreatic Elastase
Brief Title: Creon Use in Coeliac Patients With Low Faecal Pancreatic Elastase
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participant enrolment
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH16190
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Patients With Coeliac Disease and Chronic Diarrhoea (>3 Loose/ Liquid Motions a Day for More Than 4 Weeks); Patients With Pancreatic Exocrine Insufficiency
Keywords: pancreatic exocrine insufficiency; faecal elastase; diarrhoea; coeliac; creon; gastrointestinal
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Diarrhea | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Active treatment will be 2 capsules of Creon 25,000 units three times per day and the placebo will be 2 capsules three times per day; for 6 weeks treatment overall.
  Interventions: Other: Placebo
- Creon (Active Comparator): Active treatment will be 2 capsules of Creon 25,000 units three times per day and the placebo will be 2 capsules three times per day; for 6 weeks treatment overall.
  Interventions: Drug: Creon

INTERVENTIONS:
Drug: Creon — Creon is a licensed product, manufactured by Abbott Laboratories, Inc. used for the therapeutic indication of pancreatic exocrine insufficiency. The route of administration is oral, with capsules being taken with main meals without chewing. The most commonly reported adverse reactions to Creon are gastrointestinal disorders of mild or moderate severity (up to 10% of patients). These include nausea, vomiting, constipation, diarrhoea and abdominal distension. An uncommon reaction (<0.01%) of patients may develop skin reactions such as a rash or itching. No additional adverse drug reactions have been identified.
  Arms: Creon
Other: Placebo
  Arms: Placebo

SUMMARY:
Faecal elastase is an enzyme test used to identify the presence of pancreatic exocrine insufficiency. This condition manifests with symptoms of diarrhea, weight loss, causing potential impairment on an individual's quality of life. Creon, a pancreatic enzyme supplement, marketed by Abbott Laboratories, Inc. is currently the standard treatment for this condition. However, there has been limited work evaluating the merits of this medication in this condition. This study aims to evaluate the benefits that Creon may have in coeliac patients with low faecal pancreatic elastase by randomising patients with low faecal pancreatic elastase (<200 ug/g) to either treatment with Creon or placebo. Outcome measures that we aim to assess to determine the benefits of Creon include evaluation of stool frequency, abdominal pain, body mass index (BMI) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients with coeliac disease and having chronic diarrhoea (>3 loose/ liquid motions a day for more than 4 weeks)
* Patients with a low faecal elastase (<200 ug/g),
* Patients aged 16 years or over
* Patient able to give written consent to participate
* Patient not currently on Creon

Exclusion Criteria:

* Patients with normal faecal elastase (> 201ug/g),
* Patients under the age of 16
* Patients allergic to pork or any pig product (advice from the drug manufacturer)
* Patients that are pregnant or are breast-feeding
* Patients taking alternative medication that could affect bowel frequency
* Where an alternative diagnosis for the chronic diarrhoea is established, these patients will be excluded from the trial
* Patients who are unable to speak or understand English

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Stool frequency in patients with low faecal pancreatic elastase following six weeks of treatment | 6 weeks

SECONDARY OUTCOMES:
Quality of life | 6 weeks
  Quality of life on gastrointestinal symptoms in patients with low faecal pancreatic elastase following six weeks of treatment
body mass index | 6 weeks
  body mass index on gastrointestinal symptoms in patients with low faecal pancreatic elastase following six weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David S Sanders, FRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Department of Gastroenterology, Sheffield, South Yorkshire, United Kingdom